CLINICAL TRIAL: NCT04014075
Title: A Phase 2, Open-label, Single-arm Trial of Trastuzumab Deruxtecan (DS 8201a) in HER2-positive, Unresectable or Metastatic Gastric or Gastro-esophageal Junction (GEJ) Adenocarcinoma Subjects Who Have Progressed on or After a Trastuzumab-containing Regimen (DESTINY-Gastric02)
Brief Title: DS-8201a in HER2-positive Gastric Cancer That Cannot Be Surgically Removed or Has Spread (DESTINY-Gastric02)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-U205; 2019-001512-34 (EudraCT Number)
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Adenocarcinoma Gastric Stage IV With Metastases; Adenocarcinoma - GEJ
Keywords: Human epidermal receptor 2 positive; Unresectable or metastatic; HER2; Prior treatment regimen included trastuzumab
MeSH Terms: conditions — Neoplasm Metastasis | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): Participants who have centrally confirmed HER2-positive gastric or gastro-esophageal junction cancer will be treated with trastuzumab deruxtecan by intravenous (IV) infusion every 3 weeks, until progression of disease or withdrawal from treatment for other reasons.
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Antibody component covalently conjugated to a drug component, prepared by dilution based on body weight for intravenous (IV) infusion
  Other Names: DS-8201a

SUMMARY:
This study will find out if trastuzumab deruxtecan is safe and works for participants with gastric or gastroesophageal junction cancer.

They must have human epidermal growth factor receptor 2 (HER2)-positive gastric or gastro-esophageal junction (GEJ) cancer:

* that cannot be removed surgically
* that has moved to other parts of the body
* that got worse during or after treatment that included trastuzumab

The study will enroll about 80 participants. Sites will be in North America and the European Union.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years old (local regulatory guidelines apply)
* Has pathologically documented HER2-positive gastric or GEJ cancer that is unresectable or metastatic, and that progressed during or after treatment regimen containing trastuzumab
* Has at least one measurable lesion per RECIST v1.1, as confirmed by investigator review
* If of reproductive potential, agrees to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least 7 months for females and 4 months for males after the last dose of study drug

Exclusion Criteria:

* Has had anticancer therapy after first-line treatment regimen containing trastuzumab
* Has uncontrolled cardiovascular disease, including any of the following: history of myocardial infarction (MI) within 6 months of first dose or symptomatic congestive heart failure (New York Heart Association Class II to IV), troponin levels consistent with MI as defined according to the manufacturer within 28 days of first dose, or corrected QT interval (QTc) prolongation to >470 ms (females) or >450 ms (male) based on screening triplicate 12-lead electrocardiogram (ECG)
* Has history of non-infectious interstitial lung disease (ILD)/pneumonitis that required corticosteroid therapy, or current ILD/pneumonitis that cannot be ruled out at screening
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie, pulmonary emboli within 3 months of the first dose, severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive lung disease, pleural effusion, etc.), and any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (ie, rheumatoid arthritis, Sjogren's, sarcoidosis, etc.), or prior pneumonectomy.
* Has pleural effusion, ascites, or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART)
* Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms (Note: participants with clinically inactive brain metastases may be included in the study as well as participants with treated brain metastases who are no longer symptomatic and no longer require treatment with corticosteroids or anticonvulsants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (37):
- United States (20):
  - City of Hope Medical Center, Duarte, California
  - USC Norris Comprehensive Cancer Center Hospital, Los Angeles, California
  - Pacific Cancer Care, Monterey, California
  - UCLA Health, Santa Monica, California
  - Hartford Hospital, Hartford, Connecticut
  - MidState Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Miami Cancer Institute, Baptist Health South Florida, Miami, Florida
  - University of Chicago Medical Center UCMC Duchossois Center for Advanced Medicine DCAM, Chicago, Illinois
  - Kansas University Cancer Center, Kansas City, Kansas
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Alvin J. Siteman Cancer Center Washington University, St Louis, Missouri
  - Northwell Health Cancer Institute, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (3):
  - UCL St-Luc, Brussels
  - Hopital de Jolimont, Haine-Saint-Paul
  - UZ Leuven, Leuven
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Asst Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria di Modena Policlinico, Modena
  - Oncology Institute Veneto IOVIRCCS, Padua
- Spain (6):
  - Vall d'Hebron University Hospital and Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catalan de Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital la Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Biomedical Research Institute Hospital de Valencia, Valencia
- United Kingdom (4):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Royal Marsden Hospital, London
  - Christie Hospital, Manchester
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Van Cutsem E. Trastuzumab deruxtecan in HER2-positive stomach or gastroesophageal junction cancer: a plain language summary of the DESTINY-Gastric02 study. Future Oncol. 2025 Dec;21(29):3691-3700. doi: 10.1080/14796694.2025.2567230. Epub 2025 Nov 26. PMID 41294268
- [Derived] Van Cutsem E, di Bartolomeo M, Smyth E, Chau I, Park H, Siena S, Lonardi S, Wainberg ZA, Ajani J, Chao J, Janjigian Y, Qin A, Singh J, Barlaskar F, Kawaguchi Y, Ku G. Trastuzumab deruxtecan in patients in the USA and Europe with HER2-positive advanced gastric or gastroesophageal junction cancer with disease progression on or after a trastuzumab-containing regimen (DESTINY-Gastric02): primary and updated analyses from a single-arm, phase 2 study. Lancet Oncol. 2023 Jul;24(7):744-756. doi: 10.1016/S1470-2045(23)00215-2. Epub 2023 Jun 14. PMID 37329891

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 79 participants who met all inclusion criteria and no exclusion criteria were enrolled and treated at clinic centers in United States, Spain, Italy, United Kingdom, and Belgium.
Groups:
- Trastuzumab Deruxtecan: Participants who have centrally confirmed HER2-positive gastric or gastro-esophageal junction cancer received an intravenous (IV) infusion 6.4 mg/kg dose of trastuzumab deruxtecan every 3 weeks, until progression of disease or withdrawal from treatment for other reasons.
Period: Overall Study
Arm/Group | Trastuzumab Deruxtecan
Started | 79
Completed | 0
Not Completed | 79
Not completed — Progressive Disease | 53
Not completed — Adverse Event | 15
Not completed — Clinical Progression | 4
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Not completed — Miscellaneous | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Trastuzumab Deruxtecan: Participants who have centrally confirmed HER2-positive gastric or gastro-esophageal junction cancer treated with trastuzumab deruxtecan by intravenous (IV) infusion every 3 weeks, until progression of disease or withdrawal from treatment for other reasons.
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 69
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  Belgium | 4
  United States | 34
  Italy | 20
  United Kingdom | 17
  Spain | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response Rate (ORR) Based on Independent Central Review Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: The Objective Response Rate (ORR) was the defined as the percentage of participants who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), assessed by independent central review (ICR) committee based on RECIST version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Confirmed ORR based on ICR is reported.
Time Frame: Up to 16 months (data cut-off)
Population: Objective response rate was assessed in the Full Analysis Set at data cut-off date of 09 April 2021.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
Percentage of Participants | 38.0 [27.3 to 49.6]

2. Primary Outcome: Percentage of Participants With Objective Response Rate (ORR) Based on Independent Central Review Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: as for outcome 1
Time Frame: Up to 23 months (data cut-off)
Population: Objective response rate was assessed in the Full Analysis Set at data cut-off date of 08 Nov 2021.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
Percentage of Participants | 41.8 [30.8 to 53.4]

3. Secondary Outcome: Progression-Free Survival (PFS) Based on Independent Central Review Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: Progression-free survival (PFS) by independent central review was defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Up to 16 months (data cut-off)
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set at data cut-off date of 09 April 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
months | 5.5 [4.2 to 7.3]

4. Secondary Outcome: Progression-Free Survival (PFS) Based on Independent Central Review Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: as for outcome 3
Time Frame: Up to 23 months (data cut-off)
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set data at cut-off date of 08 Nov 2021
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
months | 5.6 [4.2 to 8.3]

5. Secondary Outcome: Progression-Free Survival (PFS) Based on Investigator Assessment Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: Progression-free survival (PFS) by investigator assessment was defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Up to 16 months (data cut-off)
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set at data cut-off date of 09 April 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
months | 5.5 [4.1 to 6.9]

6. Secondary Outcome: Objective Response Rate (ORR) Based on Investigator Assessment Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: The Objective Response Rate (ORR) was defined as the percentage of participants who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), assessed by investigator assessment based on RECIST version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Confirmed ORR based on investigator assessment is reported.
Time Frame: Up to 16 months (data cut-off)
Population: Objective response rate was assessed in the Full Analysis Set at data cut-off date of 09 April 2021.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
Percentage of Participants | 34.2 [23.9 to 45.7]

7. Secondary Outcome: Objective Response Rate (ORR) Based on Investigator Assessment Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: as for outcome 6
Time Frame: Up to 23 months (data cut-off)
Population: Objective response rate was assessed in the Full Analysis Set at data cut-off date of 08 Nov 2021.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
Percentage of Participants | 36.7 [26.1 to 48.3]

8. Secondary Outcome: Overall Survival (OS) Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: Overall survival (OS) was defined as the time from the date of first dose of study drug to the date of death due to any cause.
Time Frame: Up to 16 months (data cut-off)
Population: Overall survival (OS) was assessed in the Full Analysis Set at data cut-off date of 09 April 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
months | NA [11.5 to NA] — Median OS and upper limit of 95% Confidence Interval (CI) was not estimable due to insufficient number of OS events.

9. Secondary Outcome: Overall Survival (OS) Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: as for outcome 8
Time Frame: Up to 23 months (data cut-off)
Population: Overall survival (OS) was assessed in the Full Analysis Set at data cut-off date of 08 Nov 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
months | 12.1 [9.4 to 15.4]

10. Secondary Outcome: Duration of Response (DoR) Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: Duration of Response (DOR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause. DoR based on independent central review.
Time Frame: Up to 16 months (data cut-off)
Population: Duration of Response (DOR) was assessed in the Full Analysis Set at data cut-off date of 09 April 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
months | 8.1 [4.1 to NA] — The upper limit was not estimable due to the reason that the curve representing the upper confidence limits for the survivor function lies above 0.5.

11. Secondary Outcome: Duration of Response (DoR) Following Treatment With DS8201a in Participants With HER2-Positive Unresectable or Metastatic Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma
Description: as for outcome 10
Time Frame: Up to 23 months (data cut-off)
Population: Duration of Response (DOR) was assessed in the Full Analysis Set at data cut-off date of 08 Nov 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan
Number analyzed (Participants) | 79
months | 8.1 [5.9 to NA] — The upper limit was not estimable due to the reason that the curve representing the upper confidence limits for the survivor function lies above 0.5.

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up to 47 days after last dose of the study drug.
Description: A Treatment-emergent adverse event (TEAE) is defined as an AE that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the initiating the study drug until 47 days after last dose of the study drug.
Arm/Group | Trastuzumab Deruxtecan
All-Cause Mortality (participants affected / at risk) | 46/79
Serious Adverse Events (participants affected / at risk) | 37/79
Other Adverse Events (participants affected / at risk) | 79/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab Deruxtecan (N=79)
Covid-19 (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Bacterial Sepsis (Infections and infestations) | 1
Covid-19 Pneumonia (Infections and infestations) | 1
Device Related Infection (Infections and infestations) | 1
Staphylococcal Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Wound Infection (Infections and infestations) | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lymphangiosis Carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal Ganglia Infarction (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Bile Duct Stenosis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Disease Progression (General disorders) | 2
Hyperpyrexia (General disorders) | 1
Animal Bite (Injury, poisoning and procedural complications) | 1
Exposure To Communicable Disease (Injury, poisoning and procedural complications) | 1
Device Occlusion (Product Issues) | 1
Catheter Site Infection (Infections and infestations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Pyrexia (General disorders) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Deruxtecan (N=79)
Covid-19 (Infections and infestations) | 5
Device Related Infection (Infections and infestations) | 4
Anaemia (Blood and lymphatic system disorders) | 30
Neutropenia (Blood and lymphatic system disorders) | 8
Decreased Appetite (Metabolism and nutrition disorders) | 26
Hypokalaemia (Metabolism and nutrition disorders) | 13
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Insomnia (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 4
Headache (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 6
Hypotension (Vascular disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5
Nausea (Gastrointestinal disorders) | 51
Vomiting (Gastrointestinal disorders) | 35
Diarrhoea (Gastrointestinal disorders) | 29
Constipation (Gastrointestinal disorders) | 23
Abdominal Pain (Gastrointestinal disorders) | 11
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 8
Ascites (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 19
Back Pain (Musculoskeletal and connective tissue disorders) | 7
Urinary Retention (Renal and urinary disorders) | 5
Acute Kidney Injury (Renal and urinary disorders) | 4
Fatigue (General disorders) | 33
Asthenia (General disorders) | 12
Weight Decreased (Investigations) | 28
Platelet Count Decreased (Investigations) | 14
Neutrophil Count Decreased (Investigations) | 13
Aspartate Aminotransferase Increased (Investigations) | 13
White Blood Cell Count Decreased (Investigations) | 9
Alanine Aminotransferase Increased (Investigations) | 8
Blood Alkaline Phosphatase Increased (Investigations) | 9
Blood Bilirubin Increased (Investigations) | 5
Oedema Peripheral (General disorders) | 4
Urinary Tract Infection (Infections and infestations) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 4
Mucosal Inflammation (General disorders) | 4
Weight Increased (Investigations) | 5
Blood Creatinine Increased (Investigations) | 4
Pyrexia (General disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT04014075/Prot_SAP_000.pdf